CLINICAL TRIAL: NCT07192458
Title: Immunogenicity and Safety of Consecutive High-Dose vs. Standard-Dose Influenza Vaccines Administered Over Successive Seasons in Lung Transplant Recipients
Brief Title: High vs. Standard Dose Influenza Vaccines in Lung Transplant (Repeater)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Natasha Halasa, Professor of Pediatric Infectious Diseases, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 251037
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Immunization; Infection|Transplantation Infection|Influenza; Influenza
Keywords: Influenza; Vaccination; Immunization; Lung Transplantation; High Dose; Fluzone; Standard Dose; Influenza, Human; Communicable Diseases
MeSH Terms: conditions — Influenza, Human; Communicable Diseases | interventions — Influenza Vaccines; Fluzone High-Dose

STUDY DESIGN:
Intervention Model Description: The primary goal of this study is to compare influenza vaccine immunogenicity and safety between two doses of HD-QIV and two doses of SD-QIV in a population of lung transplant recipients. The study will be powered on a comparison of the primary immunogenicity outcome. A nominal level of α = 0.05 (two-sided) will be used to determine statistical significance
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study staff, and subjects will be blinded to which vaccine the subject will receive, except for an un-blinded vaccinator. This individual will not inform the study team or the subjects which vaccine they administered to the subject. The un-blinded vaccinator will not participate in any other study activities. If the study vaccine is provided in a blinded manner, then research staff will be able to administer the vaccine, and an un-blinded vaccinator will not be necessary. The pharmacy will be un-blinded and will have a record of which vaccine was given to each subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fluzone: Two Doses High Dose Inactivated Influenza Vaccine (Experimental): Fluzone: Two Doses of HD-IIV
  Interventions: Biological: Fluzone High Dose Inactivated Influenza Vaccine
- Fluzone: Two Doses Standard Dose Inactivated Influenza Vaccine (Experimental): Fluzone: Two Doses of of SD-IIV
  Interventions: Biological: Fluzone Standard Dose Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Fluzone High Dose Inactivated Influenza Vaccine — Fluzone High-Dose (Influenza Vaccine) for intramuscular use is an inactivated influenza vaccine, prepared from influenza viruses propagated in embryonated chicken eggs. The virus- containing allantoic fluid is harvested and inactivated with formaldehyde. Influenza virus is concentrated and purified in a linear sucrose density gradient solution using a continuous flow centrifuge. The virus is then chemically disrupted using a non-ionic surfactant, octylphenol ethoxylate (Triton® X-100), producing a split virus. The split virus containing hemagglutinin (HA) antigen is further purified and then suspended in sodium phosphate-buffered isotonic sodium chloride solution. The Fluzone High-Dose process uses an additional concentration factor after the ultrafiltration step to obtain a higher HA antigen concentration. The purified split virus from the three strains included in the vaccine are produced separately and then combined to make the trivalent formulation.
  Other Names: Fluzone High Dose
  Arms: Fluzone: Two Doses High Dose Inactivated Influenza Vaccine
Biological: Fluzone Standard Dose Inactivated Influenza Vaccine — Fluzone Standard Dose is a vaccine indicated for active immunization for the prevention of disease caused by influenza A subtype viruses and type B virus contained in the vaccine.
  Other Names: Fluzone
  Arms: Fluzone: Two Doses Standard Dose Inactivated Influenza Vaccine

SUMMARY:
This will be a follow-up study to the "Comparison of High Dose vs. Standard Dose Influenza Vaccine in Lung Allograft Recipient" study (DMID Protocol Number 22-0014) at Vanderbilt University Medical Center.

Lung transplantation is a life-saving therapy for patients with advanced lung disease, and is also associated with an improvement in quality of life. However, due to the need for life-long immunosuppression to prevent acute cellular rejection and chronic lung allograft dysfunction ("chronic rejection"), lung transplant recipients are at risk for developing major infections. In fact, one-year survival is 85%, with infection being the leading cause of death within the first year post-transplant. We will conduct a follow-up phase II, randomized, double-blind trial to assess the impact of subsequent administration of two doses of HD-IIV compared to two doses of SD-IIV among lung recipients during the early post-transplant period. Demonstration of improved immunogenicity from two doses of HD-IIV over consecutive influenza seasons would provide potential broad benefit in reducing influenza disease and its associated complications in lung transplant recipients. Moreover, studying vaccine immunogenicity and safety in the same participants over consecutive years can provide insight into the influence of immunosuppression levels and allograft aging on vaccine-mediated immune modulation. This proposed study design will contribute significantly to influenza vaccination guidance and policy for the highly vulnerable lung transplant population. This proposed study is designed to address several key knowledge gaps in vaccine-mediated protection of lung transplant recipients against influenza:

* Is there increased immunogenicity with administration of one or two doses of HD-IIV or SD-IIV in the subsequent season compared to two doses of HD-IIV or SD-IIV in the first season?
* What is the durability of the humoral and cellular immune response between influenza seasons and does two doses of HD-IIV or SD-IIV sustain higher HAI titers compared to two doses of HD-IIV or SD-IIV in the first season?
* What is the impact of maintenance immunosuppression levels on influenza vaccine immunogenicity within the same participant?
* Will the optimal immunogenic vaccination strategy be associated with an acceptable long-term safety profile over successive influenza seasons, including injection-site and systemic reactions, allosensitization, and organ rejection?

DETAILED DESCRIPTION:
The study is a phase II, single-center, double-blind, randomized controlled immunogenicity and safety trial comparing two doses of HD-IIV to two doses of SD-IIV over two consecutive years in lung transplant recipients. At study enrollment, following consent, participants will receive either HD-IIV or SD-IIV , with study arm assignments based on DMID protocol number 22-0014. Therefore, participants will ultimately receive four total doses of either HD-IIV or four total doses of SD-IIV over two consecutive influenza seasons.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipient who enrolled and completed Visits 1, 2, and 3 of the DMID protocol number 22-0014 during the prior 2024-2025 or 2025-2026 influenza season, respectively

  * Anticipated to be available for the duration of the study
  * Can be reached by telephone, text message, email, or electronic health record messaging

Exclusion Criteria:

* Recipient of multi-organ, extra-pulmonary, and/or hematopoietic stem cell transplant
* Recipient of a re-do lung transplant
* History of Guillain-Barre syndrome
* History of receiving the current season's influenza vaccine prior to study enrollment and/or Visit 1 of this follow-up study
* Pregnant person
* Laboratory-confirmed influenza disease after September 1st in the current influenza season and before enrollment in this follow-up study (patient can still receive the second influenza vaccination despite proven influenza disease after enrollment)
* CMVIG/IVIG/SCIG receipt within 28 days of each vaccine
* Receipt of rituximab or other B-cell depleting antibody (including proteasome inhibitors) therapy within 3 months of 1st vaccine dose (Day 0)
* Receipt of T-cell depleting therapies (anti-thymocyte globulin, alemtuzumab, daratumumab) between the completion of Visit 3 of the initial study and enrollment in this follow-up study
* Investigator concern about study participation
* Note: Criteria for temporarily delaying vaccine administration: The following conditions are temporary or self-limiting, and a participant may be included in the study once the condition has resolved, provided that the participant is otherwise eligible:

  * Fever ≥100.4ºF/38.0ºC (oral measurement), or an acute severe illness within 48 hours of enrollment
  * Receipt of any live vaccines within four weeks or any inactivated vaccines within two weeks prior to potential study vaccination

No children have been enrolled in the DMID protocol number 22-0014; therefore, only adults will be enrolled in this current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity: Geometric Mean Titers of Influenza Vaccine Antibodies | Four-eight weeks following the second study vaccination
  HAI GMT to influenza antigens four-eight weeks following the second study vaccination
Safety - The number of participants reporting solicited injection site reactions | Within 7 days post vaccination
  Solicited Injection-site Adverse Events Following each Vaccination Dose (Pain, Tenderness, Swelling/induration, Erythema/redness)
Safety - The number of participants reporting systemic adverse events | Within 7 days post vaccination
  Systemic adverse events (Fatigue/malaise, headache, nausea, body ache/myalgia (not at the injection site), general activity level, vomiting, and fever)

SECONDARY OUTCOMES:
The number of participants achieving seroprotection and seroconversion for influenza virus after receiving either two doses of HD-IIV or two doses of SD-IIV over two consecutive years | Four to eight weeks after vaccination
  Antibody titers will be measured by hemagglutination inhibition assay. Seroconversion is defined as ≥ 4-fold rise in hemagglutination inhibition assay titers. Seroprotection is defined as ≥1:40 hemagglutination inhibition assay titer.
Geometric Mean Titers of Influenza Vaccine Antibodies after One or Two Doses in the Second Year | Within four to eight weeks post vaccination after 1st and 2nd vaccine
  To quantify and compare the degree to which one versus two doses of either HD-IIV or SD-IIV in the subsequent season elicits enhanced immunogenicity compared to two doses of either HD-IIV or SD-IIV in the first influenza season in lung transplant recipients. Measuring GMT 4-8 weeks after 1st and 2nd vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Natahsa Halasa, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No